CLINICAL TRIAL: NCT03982797
Title: Treatment of High-risk Non-muscle Invasive Bladder Cancer With IMUNO BGC Moreau RJ as Prophylaxis of Recurrence and Progression.
Brief Title: Treatment of High-risk Non-muscle Invasive Bladder Cancer With IMUNO BGC Moreau RJ as Prophylaxis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biofabri, S.L (Industry)
Collaborators: Fundación para la Investigación en Urología (FIU) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENCORE-01; 2017-002928-24 (EudraCT Number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Bladder Cancer
Keywords: non-muscle invasive bladder tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated with IMUNO BCG Moreau RJ adjuvant. (Experimental)
  Interventions: Biological: Instillation of IMUNO BCG Moreau RJ

INTERVENTIONS:
Biological: Instillation of IMUNO BCG Moreau RJ — Instillation in bladder will be done once per week during first six weeks after inclusion, and 3 instillations (one per week) on month three, another three on moth six and last three on month twelve .

SUMMARY:
Bladder cancer is the fourth reason of neoplasia in our environment, there are 25 new cases diagnosed per 100,000 inhabitants each year. To decrease the recurrence there are two standardized treatments: Mitomycin as chemotherapy drug and BCG *Bacile Calmette-Guérin" as immunotherapy drug.

BCG Moreau strain is not authorized by AEMPS, it was developed in Brazil and this country has extensive experience in treatment of non-muscle invasive bladder cancer with BCG Moreau, also BCG Moreau Rio de Janeiro make same immunological reaction as TICE, but with less adverse events. Thus, BCG Moreau RJ treatment could be used more time than TICE with the same dose, keeping immunologic status and better prophylaxis of recurrence or progression results for the patient.

Each patient will be instillated via transurethral each time with 80 mg of IMUNO BCG Moreau RJ. There are 15 instillations during the clinical trial, 6 instillations on induction phase and 9 will be performed during maintaince phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the informed consent before any activity related to the study, including the necessary evaluations for the selection.
2. Age between 18 and 80 years at the time of signing the informed consent.
3. Urothelial tumor.
4. High risk non-muscle invasive bladder tumor (defined as Ta-T1 and GIIb or GIII) diagnosed de novo or relapsed with or without associated in situ carcinoma. or carcinoma in situ isolated without visible tumor.
5. Patient with risk of recurrence or progression greater than or equal to 10 points, according to CUETO tables.

Exclusion Criteria:

1. No muscle layer in pathological examination piece's.
2. Non-urothelial tumor.
3. Active cancer in any other location.
4. Diagnosis of any other pathology that in the opinion of the researcher may increase the risk of the subject or reduce the chances of obtaining satisfactory data to achieve the objectives of the study, including the consumption of alcohol or any other drug.
5. Administration of BCG in the last year before signing the informed consent. 6. BCG instillation contraindication during more than 15 days for any cause such as low bladder capacity, urinary infection, hematuria, etc.

7. Impossibility of performing a second transurethral resection (ReRTU) between 4 and 8 weeks after the first.

8. Inability to start treatment within the first 4 weeks after the second transurethral resection (ReRTU).

9. Participation in another clinical study where they received a research drug in the 6 months prior to signing the informed consent.

10. Woman considered potentially fertile. Following the Clinical Trial Facilitation Group (CTFG) recommendations, a woman is considered childbearing potential (WOCBP), following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

11. Patients with difficulties to perform the follow-up visits established in the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-04-03 (Estimated); Study Completion 2022-03-03 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 24 months
  The primary objective is to assessment the progression-free survival of patients diagnosed with high-risk non-muscle invasive bladder tumors treated with IMUNO BCG Moreau RJ adjuvant.

SECONDARY OUTCOMES:
Disease-free survival. | 24 months
  The secondary objective is to assessment the disease-free survival.
Assessment of the quality of life | 24 months
  Assessment will be measure with FACT-BL version4th
Assessment of adverse reactions | 24 months
  Assessment will be measure in number and relation with IMP
Assessment of the dropout rate due to toxicity | 24 months
  Assessment will be measure in number

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Unda, MD, Principal Investigator — Hospital Universitario Basurto
Locations (15):
- Spain (15):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Basurto, Bilbao
  - Complejo Hospitalario Puerta Del Mar, Cadiz
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Complejo Hospitalario Médico Quirúrjico de Jaén, Jaén
  - Hospital de Especialidades de Jerez de La Frontera, Jerez de la Frontera
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario Regional de Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No